CLINICAL TRIAL: NCT04481256
Title: TGF-β And PDL-1 Inhibition in Esophageal Squamous Cell Carcinoma Combined With Chemoradiation TheRapY
Acronym: TAPESTRY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other); Catharina Ziekenhuis Eindhoven (Other); Institute Verbeeten (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Leiden University Medical Center (Other); Radiotherapeutic Institute Friesland (Other); Frisius Medisch Centrum (Other); Radiotherapy Group Deventer (Other); Deventer Ziekenhuis (Other); Rijnstate Hospital (Other); Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); Isala (Other); University Medical Center Groningen (Other); Ziekenhuisgroep Twente (Other)
Responsible Party: Principal Investigator, Hanneke W. M. van Laarhoven, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73750; NCT04595149 (obsolete NCT alias)
Record Dates: First submitted 2020-05-26; First posted 2020-07-22 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Squamous Cell; Oesophageal Cancer
Keywords: Definitive chemoradiation; TGF-beta inhibition; PDL-1 ihibition; feasability
MeSH Terms: conditions — Carcinoma, Squamous Cell; Esophageal Neoplasms | interventions — bintrafusp alfa protein, human; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Non-randomized feasibility study with paclitaxel, carboplatin, bintrafusp alfa, and radiation. Paclitaxel 50 mg/m2 and carboplatin AUC = 2 will be given intravenously (i.v.) on days 1, 8, 15, 22, 29 and 36. Bintrafusp alfa will be given i.v. every three weeks on day 1, 22, and 43 at a dose of 2400 mg. External beam radiotherapy will be delivered to a total dose of 50.4 Gy in 28 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 Bintrafusp alfa, Paclitaxal, Carboplatin, Radiotherapy (Experimental): Non-randomized feasibility study with paclitaxel, carboplatin, bintrafusp alfa, and radiation. Paclitaxel 50 mg/m2 and carboplatin AUC = 2 will be given intravenously (i.v.) on days 1, 8, 15, 22, 29 and 36. Bintrafusp alfa will be given i.v. every three weeks on day 1, 22, and 43 at a dose of 2400 mg.
  External beam radiotherapy will be delivered to a total dose of 50.4 Gy in 28 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy
  Interventions: Radiation: External beam radiotherapy; Drug: Bintrafusp alfa; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: External beam radiotherapy — External beam radiotherapy will be delivered to a total dose of 50.4 Gy in 28 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy
Drug: Bintrafusp alfa — Bintrafusp alfa will be given i.v. every three weeks on day 1, 22, and 43 at a dose of 2400 mg.
  Other Names: M7824
Drug: Paclitaxel — Paclitaxel 50 mg/m2 will be given intravenously (i.v.) on days 1, 8, 15, 22, 29 and 36.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin AUC = 2 will be given intravenously (i.v.) on days 1, 8, 15, 22, 29 and 36.

SUMMARY:
The primary objective of this study is to assess the feasibility of treatment with bintrafusp alfa combined with definitive chemoradiation (carboplatin, paclitaxel and radiation) in patients with squamous cell carcinoma of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
Non-randomized feasibility study with paclitaxel, carboplatin, bintrafusp alfa, and radiation. Paclitaxel 50 mg/m2 and carboplatin AUC = 2 will be given intravenously (i.v.) on days 1, 8, 15, 22, 29 and 36. Bintrafusp alfa will be given i.v. every three weeks on day 1, 22, and 43 at a dose of 2400 mg. External beam radiotherapy will be delivered to a total dose of 50.4 Gy in 28 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the esophagus or gastro esophageal junction.
* Surgically irresectable (T1-T4a, N0 or N+, M0), as determined by Endoscopic Ultra Sound (EUS), PET scan and diagnostic CT scan of neck, thorax and abdomen. Patients with M1 disease solely on the basis of supraclavicular metastasis are eligible. Patients with resectable tumors refusing radical surgery are eligible.
* Locoregional recurrences without distant metastasis after surgery alone or endoscopical resection
* Locoregional recurrences without distant metastasis after neoadjuvant chemoradiation + resection or definitive chemoradiation outside the previously irradiated area, provided that full dose of radiation can safely be delivered.
* Tumors that cannot be passed with an endoscope for endoscopic ultrasound are eligible if all other criteria are fulfilled.
* If the tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction.
* Age ≥ 18.
* ECOG performance status 0-2 (cf. Appendix A).
* Adequate hematological, renal and hepatic functions defined as:

  * Neutrophils ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 5.6 mmol
  * Total bilirubin ≤ 1.5 x upper normal limit
  * ASAT and ALAT ≤ 1.5 x upper normal limit, Alkaline Phosphatase ≤ 2.5 x upper normal limit.
  * PT (INR) ≤ 1.5 x upper normal limit and aPTT ≤ 1.5 x upper normal limit.
  * Creatinine clearance (Cockroft) > 60 ml/min
* Written, voluntary informed consent
* Patients must be accessible to management and follow-up in the treatment center

Exclusion Criteria:

* Past or current history of malignancy other than entry diagnosis interfering with prognosis of esophageal cancer.
* Patient with tracheo-esophageal fistula or extension into the mucosal layer of the trachea, highly at risk to develop fistula. Thus, tumor extension to the trachea is allowed, but not through the trachea.
* Patients with pathological lymph nodes at both supraclavicular and truncus coeliacus level.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Patient (male or female) in the reproductive age is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Previous chemotherapy, radiation and/or treatment with checkpoint inhibitors for the currently present esophageal tumor.
* Previous chemotherapy and/or treatment with targeted agents and/or checkpoint inhibitors for other forms of cancer within the last six months.
* Previous radiation to the mediastinum precluding full dose radiation of the currently present esophageal tumor.
* Persisting grade >1 NCI CTCAE 5.0 toxicity (except alopecia and vitiligo) related to prior therapy; however, grade ≤2 sensory neuropathy is acceptable.
* Presence of an esophageal stent.
* History of bleeding diathesis or major bleeding event (grade ≥ 2) in the month prior to first dose of trial treatment.
* Current use of direct oral anticoagulants or coumarins.
* Clinically significant cardiovascular disease precluding safe treatment with chemoradiation.
* Evidence of pulmonary fibrosis and/or clinically significant impairment of lung function precluding safe treatment with chemoradiation. In case of doubt about pulmonary function, a lung function test should be performed and, in case of abnormalities, discussed with the principle investigator.
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing cremophor, such as teniposide or cyclosporine.
* Mental status that would prohibit the understanding and giving of informed consent.
* Inadequate caloric- and/or fluid intake despite consultation of a dietician and/or tube feeding.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine for patients with a history of autoimmune-related hypothyroidism, insulin for patients with type 1 diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo with dermatological manifestations only are eligible to enter the study.
* A diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Diagnosis of HIV unless stable on antiretroviral therapy for at least 4 weeks, no evidence of multi-drug resistance, viral load of < 400 copies/ml and CD4+ T-cells ≥ 350 cells/µl.
* Active HBV/HCV. Participants on a stable dose of antiviral therapy with HBV/HCV viral load below the limit of quantification are eligible.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* An active infection requiring systemic therapy, which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Administration of a live vaccine within 30 days prior to the first dose of trial treatment. Seasonal flu vaccines that do not contain a live virus are permitted.
* Patients with prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility difined as the percentage of patients completing at least two cycles of bintrafusp alfa | 36 months
  The primary outcome of this study is the percentage of patients that completes at least two cycles of bintrafusp alfa together with their chemoradiotherapy regimen.

SECONDARY OUTCOMES:
Incidence and severity of toxicity | 36 months
  Incidence and severity of toxicity defined according to CTCAE v5 and and Radiation Oncology Group (RTOG) criteria.
Percentage completion | 36 months
  Percentage completion of chemotherapy and radiation treatment
Percentage withdrawal rate | 36 months
  Percentage withdrawal rate from chemoradiation due to bintrafusp alfa related complications
locoregional progression | 36 months
  Infield locoregional progression free survival
progression | 36 months
  Any progression free survival
Survival | 36 months
  Overall survival
Quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ C30)) | 36 months
  Overall Quality of life ranging from 0-100 with 100 being best Quality of Life with special focus on dysphagia
adverse events | 36 months
  To determine the number and grade of adverse events of bintrafusp alfa combined with chemoradiotherapy according to NCI common toxicity criteria (CTC) version 5

OTHER OUTCOMES:
Biomarker | 54 months
  To perform exploratory biomarker analyses for treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, MD,PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No